CLINICAL TRIAL: NCT07087938
Title: Safety and Behavioral Pharmacology of Cannabichromene as an Adjunct to Rheumatoid Arthritis Treatment; Effects on Inflammatory Markers and Rheumatoid Arthritis Disease Activity
Brief Title: Cannabichromene Safety in Rheumatoid Arthritis
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was put on clinical hold with the FDA prior to beginning enrollment due to insufficient preclinical evidence.
Sponsor: Crystal Lederhos Smith (Other)
Responsible Party: Sponsor-Investigator, Crystal Lederhos Smith, Assistant Professor, Washington State University
Organization: Washington State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20353-001
Record Dates: First submitted 2024-05-31; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Cannabichromene; CBCH; CBC; Minor cannabinoid; CBC in humans; Rheumatoid Arthritis; Safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cannabichromene

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to begin with one of two study doses (400mg or 600mg daily) using a block randomization schedule.
Who Masked: Participant
Masking Description: Participants will be blinded to dose but will know they are all getting active product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group 1 (Active Comparator): Participants will be administered dose one (400mg CBC daily) for eight weeks, and at visit three they will receive dose two (600mg CBC daily) and will take it for eight weeks, concluding the study with another two-week washout period.
  Interventions: Drug: Cannabichromene
- Study Group 2 (Active Comparator): Participants will be administered dose one (600mg CBC daily) for eight weeks, and at visit three they will receive dose two (400mg CBC daily) and will take it for eight weeks, concluding the study with another two-week washout period.
  Interventions: Drug: Cannabichromene

INTERVENTIONS:
Drug: Cannabichromene — Participants will be assigned (using block randomization) to begin with one of the two study doses of CBC (400mg or 600mg). Participants will be blinded to dose. They will be asked to take half of their dose in the morning and half in the evening. Participants will be administered dose one for eight weeks. After this, participants will have a two-week timeframe where they will be asked not to take any study medication and to continue refraining from cannabis use, thus providing a washout period. Then, at visit three, they will receive dose two and will take it for eight weeks, concluding the study with another two-week washout period. At each clinic visit participants will complete assessments (self-report and physical examination), urine, and blood samples.
  Other Names: CAS Number: 20675-51-8; CBC; NSC 291831

SUMMARY:
For this quantitative study, the investigators will collect data on human safety and side-effects of Cannabichromene (CBC) and whether CBC reduces blood inflammatory markers and Rheumatoid Arthritis (RA) disease activity. The participants will participate in an ABAB design with 2 doses of CBC across the A phases. They will attend 5 in-person clinic visits where they will have physical evaluations, complete self-report forms, and have blood drawn for the following tests: hs-CRP, ESR, IL-6, TNF, Complete Blood Count [CBC], and CMP.

DETAILED DESCRIPTION:
Due to their anti-inflammatory effects, cannabinoids have been considered as a potential therapy for the treatment of rheumatic diseases in humans. However, there is not yet significant evidence for the efficacy of cannabinoid-based treatments for rheumatoid arthritis, even though it is included in the list of eligible conditions for medical cannabis in Canada and many US states. In this study, the investigators propose to examine the safety and human behavioral pharmacology of CBC:

No statistical hypotheses have been developed for Aims 1 and 2 as they are descriptive in nature. Aim 3 has the statistical hypothesis embedded within it. These are reiterated below:

Aim 1: Assess human safety of CBC through a count of the number of treatment-related adverse events experienced by participants. This is a descriptive aim and therefore does not have an associated hypothesis.

Aim 2: Assess human safety of CBC through measurement of blood markers indicating organ function. This is a descriptive aim wherein the investigators will provide a qualitative description of changes in blood markers during treatment; it therefore does not have an associated hypothesis.

Aim 3: Determine if CBC reduces blood inflammatory markers and overall rheumatoid arthritis disease activity (as measured by the DAS28), across 2 dosages (400mg and 600mg CBC daily), each administered for an 8-week period. The investigators hypothesize that CBC will yield lower levels of inflammatory markers and overall disease activity during the treatment period and that levels of inflammatory markers will return to baseline at the 2-week follow-up for both of the doses.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of RA
* Having stable treatment for at least 1 month prior to the study and being willing to continue that treatment for the duration of the study
* Having some degree of disease activity present at research study intake (determined by research study personnel)
* Aged 21+
* Able to read and speak English, and provide written consent
* Not currently pregnant or planning to become pregnant during the trial
* Not currently planning any surgeries during the course of the trial
* Willing to use a form of birth control for the duration of the study (all participants will be required to use birth control for the duration of the study)
* Willing to refrain from cannabis use (other than study provided CBC) over the course of the study

Exclusion Criteria:

* Do not have a current diagnosis of RA
* Has not received stable treatment for at least 1 month prior to the study or is unwilling to continue treatment for the duration of the study
* No degree of disease activity present at research study intake (determined by research study personnel)
* Under age 21
* Unable to read and speak English, or provide written consent
* Are currently pregnant or planning to become pregnant during the course of the trial
* Unwilling to use a form of birth control during the duration of the study
* Is planning a surgery during the course of their participation in the trial
* Unwilling to refrain from cannabis use (other than study provided CBC) over the course of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2028-07-15 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Observed Adverse Events | 20 Weeks
  Observed Adverse events
Incidence of Serious Adverse Events | 20 Weeks
  Observed Serious adverse events
Incidence of Side-Effects Reported by Participants | 20 Weeks
  Participant self-report of side-effects
Description of Safety Focused Blood Markers (CMP) | 20 Weeks
  Safety focused blood marker levels aggregated through Comprehensive Metabolic Panel (CMP) during the treatment and post treatment phases.
Description of Safety Focused Blood Markers (CBC) | 20 Weeks
  Safety focused blood marker levels aggregated through Complete Blood Count (CBC) during the treatment and post treatment phases.

SECONDARY OUTCOMES:
Number of Participants With CBC Treatment-Related Reduction of RA Disease Activity as Assessed by DAS28. | 20 Weeks
  Overall Rheumatoid Arthritis disease activity as assessed by the DAS28 (Disease Activity Score in 28 joints) tool across 2 dosages (400mg and 600mg daily), administered for 8 weeks per dose.
Number of Participants With CBC Treatment-Related Reduced Inflammatory Blood Markers as Assessed by hs-CRP, ESR, IL-6, and TNF Tests. | 20 Weeks
  This will be measured across 2 dosages (400mg and 600mg daily), administered for 8 weeks per dose.
  This will be determined through the collection of inflammation focused blood marker levels during the treatment and post treatment phases: (High sensitivity C-reactive protein (hs-CRP); Erythrocyte Sedimentation Rate (ESR); Interleukin-6 (IL-6); Tumor Necrosis Factor (TNF) )

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Smith, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified and summarized participant data will be available to other researchers upon request. No IPD will be available due to the focused recruitment strategy, in an effort to provide protection to participants identities.